CLINICAL TRIAL: NCT00717639
Title: Determination of Diagnostic Accuracy and Added Value of Vasovist®-Enhanced Peripheral MRA in Comparison to Intra-arterial Digital Subtraction Angiography (i.a. DSA) in Patients With Peripheral Artery Disease
Brief Title: Vasovist Magnetic Resonance Angiography (MRA) in Peripheral Arterial Occlusive Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Required contrast media (Vasovist) withdrawn from market
Sponsor: Heidelberg University (Other)
Responsible Party: Henrik Michaely (Principal Investigator), University of Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Vasovist MA-01; EudraCT 2007-006014-41
Record Dates: First submitted 2008-06-30; First posted 2008-07-17 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2010-07

CONDITIONS: Peripheral Arterial Occlusive Disease
Keywords: diagnostic accuracy; magnetic resonance angiography; steady state; digital subtraction angiography; peripheral arteries
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): single arm study, all patients will undergo Vasovist-enhanced MRA
  Interventions: Procedure: Diagnostic MR-Angiography

INTERVENTIONS:
Procedure: Diagnostic MR-Angiography — Single MR-Angiography of the lower extremity after the bolus injection 0.03mmol/kg BW Vasovist
  Other Names: Vasovist(R); generic name - gadofosveset

SUMMARY:
This study aims at investigating the diagnostic accuracy of magnetic resonance angiography using the contrast agent Vasovist® in the detection of relevant vascular narrowing of the lower extremity. Patients who have been scheduled for intra-arterial conventional angiography are eligible for this trial.

DETAILED DESCRIPTION:
Patients will only be included into the study if either MRA with extracellular contrast agents, computed tomography angiography, ultrasound or i.a. DSA have been performed beforehand and if the patient has been scheduled for an i.a. DSA to be performed. Vasovist® enhanced MRA imaging will be performed using a state-of-the-art 1.5T MR system. Recruitment, baseline examinations, Vasovist®-enhanced MRA of the vessel segments of interest and follow-up examinations will be performed in up to 8 radiological clinics in Europe. The safety follow-up period will be at least 12 hours but not more than 24 hours post injection of Vasovist® and includes the assessment of physical examinations and vital signs as well as the assessment of AEs. DSA must be carried out at least 12 hours after Vasovist® administration and only after the last follow-up visit has been performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have Fontaine-stage III and IV and an indication for therapeutic i.a. DSA
* PAOD has to be confirmed by ECCM MRA, CTA, non-selective DSA, Doppler ultrasound (DUS) prior to the study.
* Patients who are willing to undergo the study MRA procedure with Vasovist
* Patients who are willing to comply with the study procedures (e.g. being followed-up for 12 hours after the Vasovist injection).
* Patients who have given their fully informed and written consent voluntarily.

Exclusion Criteria:

* Being less than 18 years of age.
* Women who are pregnant, lactating or who are of childbearing potential and have not had a negative urine pregnancy test the same day as administration of Vasovist. The manufacturer's instructions for performing the urinary pregnancy test are to be followed.
* Patients who are scheduled for any therapy between any of the two procedures (MRA and DSA) that interferes with the comparability of the two angiographic procedures.
* Having an underlying disease or concomitant medication which may interfere with efficacy or safety evaluations as planned in this study.
* Having any physical or mental status that interferes with the informed consent procedure including self-signed consent.
* GFR < 30 ml/m²/1.73m² (MDRD), values ≤ 1 week or patients on hemodialysis
* Renal or liver transplant patients, including patients with scheduled liver transplant are excluded due to the potential risk for nephrogenic systemic fibrosis (NSF).
* MR contraindications (pacemaker, magnetic clips, severe claustrophobia)
* Known allergy to Gadofosveset
* Presenting with history of anaphylactoid or anaphylactic reaction to any allergen including drugs and contrast agents.
* Untreated significant stenosis in pelvis
* Known severe coagulopathy (PTT > 25s, Quick < 60%)
* Having received any investigational drug within 7 days prior to entering this study or who are planned to receive any investigational drug during the safety follow-up period.
* Not being able to remain lying down for at least 30-45 min (e.g. patients with unstable angina, dyspnea at rest, severe pain at rest, severe back pain).
* Being clinically unstable and whose clinical course during the 12 hours observation period is unpredictable.
* Being scheduled for, or likely to require, any surgical intervention within 12 hours before or within the follow-up period.
* Patients in whom i.a. DSA is contra-indicated preventing him/her from undergoing standard of reference (SOR) procedure.
* Close affiliation with the investigational site; e.g. a close relative of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Accuracy of quantitative stenosis grading (<50%, >=50%) of Vasovist enhanced MRA with regard to i.a. DSA as standard of reference | End of study (anticipated Sep 2009)

SECONDARY OUTCOMES:
Proportion of correct stenosis gradings (<50%, 50-99%, occlusion) of Vasovist® enhanced MRA compared to DSA | End of study
Sensitivity and specificity (<50%, >=50%) of Vasovist enhanced MRA compared to DSA | End of study
Length of stenosis (target) of Vasovist® enhanced MRA compared to DSA | End of study
Correlation of the description of the inflow, target, outflow of Vasovist® enhanced MRA (combined) compared to DSA | End of study
Diagnostic value (detection of target lesion y/n) of time-resolved first pass MRA in comparison to high-spatial resolution steady state MRA | End of study
Additional venous pathologies | End of study
Diagnostic confidence of Vasovist enhanced MRA and DSA | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Henrik J Michaely, MD, Principal Investigator — Heidelberg University; Stefan O Schoenberg, MD, Study Director — Heidelberg University
Locations (2):
- Germany (2):
  - University Medical Center Mannheim, Mannheim
  - University of Munich, Munich